CLINICAL TRIAL: NCT01680653
Title: Pilot Study in Testing State of the Art Remote Glucose Monitoring at Diabetes Camp
Brief Title: Testing State of the Art Remote Glucose Monitoring at Diabetes Camp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Virginia (Other); DexCom, Inc. (Industry); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Principle Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012PG-T1D001; IRB 27428 (Other: Stanford IRB)
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2017-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon; Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mini-Glucagon and Remote Monitoring (Experimental): Subjects glucose data are remotely monitored at night using the University of Virginia (UVA) Diabetes Assistant (DiAs) Android Platform. Study staff intervenes with a fingerstick blood glucose measurement when sensor value falls below 70mg/dL. If fingerstick value is less than 70 mg/dL, hypoglycemic treatment is administered as below.
  Administer mini-glucagon as treatment for nocturnal hypoglycemia. Administer 0.01 cc per number of years in age via insulin syringe, subcutaneously. This amounts to 1 unit per age, for example: an 8 year old gets 8 "units" glucagon.
  Interventions: Drug: Mini-glucagon; Device: Remote monitoring
- Carbohydrates and Remote Monitoring (Other): Subjects glucose data are remotely monitored at night using the University of Virginia (UVA) Diabetes Assistant (DiAs) Android Platform. Study staff intervenes with a fingerstick blood glucose measurement when sensor value falls below 70mg/dL. If fingerstick value is less than 70 mg/dL, hypoglycemic treatment is administered as below.
  Administration of carbohydrate per camp protocol to treat nocturnal hypoglycemia. Expected treatment is 15-45g.
  Interventions: Device: Remote monitoring; Dietary Supplement: Carbohydrates
- Carbohydrates No Remote Monitoring (Other): Subjects wear a continuous glucose monitor for their own use, but they are not remotely monitored.
  If hypoglycemia occurs and is acknowledged through standard camp protocol it will be treated with standard camp protocol administration of carbohydrates. Expected treatment is 15g-45g.
  Interventions: Dietary Supplement: Carbohydrates
- Mini-Glucagon and No Remote Monitoring (Other): Subjects wear a continuous glucose monitor for their own use, but they are not remotely monitored.
  If hypoglycemia occurs and is acknowledged through standard camp protocol it will be treated with mini-glucagon.
  Administer mini-glucagon as treatment for nocturnal hypoglycemia. Administer 0.01 cc per number of years in age via insulin syringe, subcutaneously. This amounts to 1 unit per age, for example: an 8 year old gets 8 "units" glucagon.
  Interventions: Drug: Mini-glucagon

INTERVENTIONS:
Drug: Mini-glucagon — Mini dose glucagon given for glucose <70 mg/dl at a dose of 1unit/year of age
  Other Names: glucagon
  Arms: Mini-Glucagon and No Remote Monitoring; Mini-Glucagon and Remote Monitoring
Device: Remote monitoring — Provides real-time continuous glucose monitoring
  Arms: Carbohydrates and Remote Monitoring; Mini-Glucagon and Remote Monitoring
Dietary Supplement: Carbohydrates — 16 grams of carbohydrate
  Arms: Carbohydrates No Remote Monitoring; Carbohydrates and Remote Monitoring

SUMMARY:
The incidence of low blood sugar and hypoglycemic seizures at diabetes camp has been reduced thanks to overnight blood glucose level testing. The timing of the overnight blood test is often arbitrary and it is unclear when the highest frequency of nocturnal hypoglycemic events at camp are occurring. It is also unclear what the most appropriate treatment for nocturnal hypoglycemia is: simple carbohydrates, or mini-glucagon.

In this study, we will use Continuous Glucose Monitors (CGMs) that will send subject data securely to a remote computer located in the medical cottage at camp throughout the night. Study staff will monitor the computer and will intervene on low blood sugar as it occurs in real time. On half of the nights, campers will receive mini-glucagon for low blood sugar, and on the rest, they will receive standard carbohydrate treatment.

DETAILED DESCRIPTION:
The study will include approximately 20 subjects with Type 1 Diabetes per camp session. 10 will be linked to remote monitoring with the Diabetes Assistant Computational/Communication platform (DIAs), and 10 will wear the Dexcom CGM with the same threshold alarm setting as those wearing the DiAs (70 mg/dl), but without remote monitoring.

Study participants will be between the ages of 7-21 with type 1 diabetes. This would allow for a counselor in training or a young counselor with a history of recent nocturnal hypoglycemia to be included. It is these late adolescents and young adults who often have the most severe hypoglycemic events during a camp session. We will preferentially recruit campers into the study who: 1) have a history of nocturnal hypoglycemia requiring treatment within the last 2 months, 2) have hypoglycemia unawareness confirmed with the Clark screening test, 3) have an A1c of <8% while requiring >0.7 units/kg/day of insulin and diabetes duration of > 1year.

At the beginning of camp, a Dexcom G4 sensor will be inserted into each participating subject and after the initial calibration, they will be calibrated with blood glucose levels in the morning and before bed each day as well as when the Dexcom sensor requests a calibration. All insulin doses and treatment decisions at camp will be based on capillary blood glucose levels and they will not be based on sensor readings. Each night, 10 of the 20 campers will be randomly assigned to remote monitoring. The randomization schedule will be computer generated prior to camp. A hypoglycemia threshold will be set for 70 mg/dl. The Dexcom communicating with the DiAs will not sound a local alarm, but an alarm will be generated at the remote monitoring. Medical personnel on call at the remote monitoring station will come to the camper's cabin and confirmatory capillary blood glucose (CBG) glucose will be obtained. If the camper is <70 hypoglycemia, treatment will be given (we will not use predictive alarms or use the rate of change to determine treatment). Treatment will be randomized to mini-glucagon or standard oral treatment if campers are <70 mg/dl in a 1:1 ratio. All subjects less than 70 mg/dl will then be retested in 15 minutes with a CBG to confirm recovery from hypoglycemia.

If a sensor should fail or be dislodged during camp, it will be replaced. If a sensor needs to be replaced more than 2 times, a subject may be dropped and a different subject enrolled.

There will be a designed medical staff person who will be monitoring subjects remotely each night. A second staff person will be available to go to subjects cabins to provide treatment for hypoglycemia. If a second event should occur at the same time, a third staff person will be "on call" to attend the second camper.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year
* Age 7-21 years
* Attendee of Camp De Los Ninos or Conrad Chinnock
* Come to camp with a consent already signed after having talked to study staff about the study, or at the onset of the camp meet with study staff and sign the consent before the first night at camp.
* Using multiple daily insulin injections (Lantus) or on an insulin pump (any brand)

Exclusion Criteria:

* Cystic fibrosis
* Medications such as current use of oral steroids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* History of adhesive allergies which would interfere with sensor wear.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] DeSalvo DJ, Keith-Hynes P, Peyser T, Place J, Caswell K, Wilson DM, Harris B, Clinton P, Kovatchev B, Buckingham BA. Remote glucose monitoring in camp setting reduces the risk of prolonged nocturnal hypoglycemia. Diabetes Technol Ther. 2014 Jan;16(1):1-7. doi: 10.1089/dia.2013.0139. Epub 2013 Oct 29. PMID 24168317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were recruited from clinic; if more than 20 subjects were interested in participating in a given session, we preferentially enrolled those with a history of nocturnal awareness confirmed within the previous 2 months, (hypoglycemia unawareness confirmed with the Clarke screening test), or A1c <8% needing >0.7 units/kg day insulin.
Groups:
- All Participants: The subjects participated in three camps; each camp had approximately 20 subjects. There were two locations, one hosting two sessions. Each camp was approximately 5-6 days in length. Campers wore the device on alternating days, and hypoglycemia was treated with either mini glucagon or carbohydrates.
Period: Overall Study
Arm/Group | All Participants
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: The subjects were enrolled at three camps for diabetes; from each camp approximately 20 subjects were enrolled. There were two locations, one hosting two sessions. Each camp was approximately 5-6 days in length. Campers wore a continuous glucose sensor every day they were in the study. On alternate nights they had remote monitoring, this defined the primary treatment arms: remote monitoring or no remote monitoring. On alternating days of remote monitoring hypoglycemia was treated with either mini glucagon or carbohydrates, this was a secondary randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (3.8)
Age, Customized [Count of Participants; unit: Participants]
  7-11 years | 12
  12-16 years | 39
  17-21 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 39
  More than one race | 0
  Unknown or Not Reported | 18
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Duration of Nocturnal Hypoglycemia
Description: Number of minutes with glucose reading < 50 mg/dL. Each camper had Remote Monitoring nights and Control nights.
Time Frame: 8 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: Hypoglycemic events
Groups:
- Remote Monitoring: Subjects glucose data are remotely monitored at night using the University of Virginia (UVA) Diabetes Assistant (DiAs) Android Platform. Study staff intervenes with a fingerstick blood glucose measurement when sensor value falls below 70mg/dL. If fingerstick value is less than 70 mg/dL, hypoglycemic treatment is administered as below.
  Administer mini-glucagon as treatment for nocturnal hypoglycemia. Administer 0.01 cc per number of years in age via insulin syringe, subcutaneously. This amounts to 1 unit per age, for example: an 8 year old gets 8 "units" glucagon.
  Mini-glucagon: Mini dose glucagon given for glucose <70 mg/dl at a dose of 1unit/year of age
  Remote monitoring: Provides real-time continuous glucose monitoring
- Control: Subjects glucose data are remotely monitored at night using the University of Virginia (UVA) Diabetes Assistant (DiAs) Android Platform. Study staff intervenes with a fingerstick blood glucose measurement when sensor value falls below 70mg/dL. If fingerstick value is less than 70 mg/dL, hypoglycemic treatment is administered as below.
  Administration of carbohydrate per camp protocol to treat nocturnal hypoglycemia. Expected treatment is 15-45g.
  Remote monitoring: Provides real-time continuous glucose monitoring
  Carbohydrates and remote monitoring: 16 grams of carbohydrate with remote monitoring
Arm/Group | Remote Monitoring | Control
Number analyzed (Participants) | 57 | 57
Number analyzed (Hypoglycemic events) | 24 | 41
minutes | 12.5 [10 to 20] | 15 [10 to 30]
Statistical Analysis 1: Comparison: Remote Monitoring vs Control; The study was a feasibility and preliminary safety study. As such, the sample size was not statistically derived and the protocol was not powered to provide for definitive conclusions. The study was limited to 20 participants at each camp session. A hypoglycemic event was defined as at least two consecutive CGM readings (10 mins) below the hypoglycemic threshold of <70 mg/dL. Recovery from a hypoglycemic event required readings above threshold for > or = 25 minutes; Test type: Superiority or Other; p = 0.106, Wilcoxon (Mann-Whitney) — In analyzing prolonged events on remote monitoring versus control, we used x squared analysis or Fisher's exact test to analyze data on 2 x 2 contingency tables. Significance was defined as P<0.05

2. Secondary Outcome: Duration of Glucose Readings <70 mg/dl
Description: Number of minutes with glucose reading < 70 mg/dL. Each camper had Remote Monitoring nights and Control nights.
Time Frame: 8 Hours
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: Hypoglycemic events
Groups:
- Remote Monitoring: Subjects glucose data are remotely monitored at night using the University of Virginia (UVA) Diabetes Assistant (DiAs) Android Platform. Study staff intervenes with a fingerstick blood glucose measurement when sensor value falls below 70mg/dL. If fingerstick value is less than 70 mg/dL, hypoglycemic treatment is administered as below.
  Remote monitoring: Provides real-time continuous glucose monitoring
- Control (no Remote Monitoring): Subjects glucose data are remotely monitored at night using the University of Virginia (UVA) Diabetes Assistant (DiAs) Android Platform. Study staff intervenes with a fingerstick blood glucose measurement when sensor value falls below 70mg/dL. If fingerstick value is less than 70 mg/dL, hypoglycemic treatment is administered as below.
Arm/Group | Remote Monitoring | Control (no Remote Monitoring)
Number analyzed (Participants) | 57 | 57
Number analyzed (Hypoglycemic events) | 78 | 119
minutes | 30 [20 to 45] | 35 [25 to 72.5]
Statistical Analysis 1: Comparison: Remote Monitoring vs Control (no Remote Monitoring); Test type: Superiority or Other; p = 0.078, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Prolonged Episodes of Hypoglycemic Events
Description: Prolonged hypoglycemia is defined as glucose readings of either <70 mg/dL for greater than one hour on and off the device, <70 mg/dL for greater than 2 hours on and off the device, <50 mg/dL that lasted longer than 30 minutes on and off the device and readings of <50 mg/dL for longer than an hour, again for both the control and the subjects that were remotely monitored with the device. Each camper had Remote Monitoring nights and Control nights.
Time Frame: 8 hours at night
Measure: Number; unit: events
Groups:
- Remote Monitoring: Subjects who were on the device during the night (remotely monitored)
- Control: Subjects who were not being remotely monitored (not on the device)
Arm/Group | Remote Monitoring | Control
Number analyzed (Participants) | 57 | 57
events
  Events <70 mg/dL >1 hour | 7 | 33
  Events <70 mg/dL >2hr | 0 | 12
  Events <50 mg/dL >30 mins | 0 | 9
  Events <50 mg/dL >1hr | 0 | 6
Statistical Analysis 1: Comparison: Remote Monitoring vs Control; This is the P value for the number of events <70 mg/dL longer than one hour; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney); Fisher's exact test
Statistical Analysis 2: Comparison: Remote Monitoring vs Control; This is the p value for the number of events <70 mg/dL that were greater than 2 hours; Test type: Superiority or Other; p = 0.010, Fisher's exact test
Statistical Analysis 3: Comparison: Remote Monitoring vs Control; This is the p value for the number of events that were <50 mg/dL for > 30 minutes; Test type: Superiority or Other; p = 0.021, Fisher's exact test
Statistical Analysis 4: Comparison: Remote Monitoring vs Control; This is the P value for the number of events <50 mg/dL that were >1 hr; Test type: Superiority or Other; p = 0.077, Fisher's exact

ADVERSE EVENTS:
Time Frame: AE data was collected during the camp study periods (from 5-6 days for each of the 3 camps).
Description: Serious hypoglycemic events are recorded as AEs if the event required assistance due to altered consciousness and required another person to actively administer treatment. Hyperglycemic events are AEs if the event involved DKA, polyuria, polydipsia, nausea, vomiting, serum ketones, blood pH <7.3, venous pH <7.24, or serum bicarbonate <15
Groups:
- Remote Monitoring; Control (no Remote Monitoring): All participants; during the study, each subject was randomized to either the control or the remote monitoring group, and then alternated on subsequent nights.
Arm/Group | Remote Monitoring | Control (no Remote Monitoring)
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 3/57 | 3/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote Monitoring (N=57) | Control (no Remote Monitoring) (N=57)
mild erythema from the adhesive (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) — 5% of the campers had mild erythema from the adhesive, and there was no significant edema or induction at the sensor insertion sites.

LIMITATIONS AND CAVEATS:
Limitations revolved around sensor failure. There was one subject removed because of improper use of the device (turning it off at improper times and failing to calibrate as instructed).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No